CLINICAL TRIAL: NCT00197288
Title: A Phase III, Observer-blind, Randomized Study to Evaluate the Immunogenicity and Safety of Fluarix™ (GlaxoSmithKline Biologicals) Compared With Fluzone® (Aventis Pasteur) Administered Intramuscularly in Adults 18 Years and Older in the U.S.
Brief Title: Study Comparing the Immune Response of Fluarix and Fluzone Influenza Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 104437
Record Dates: First submitted 2005-09-19; First posted 2005-09-20 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Influenza
Keywords: Prophylaxis: Influenza virus infection
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Biological: Influenza

SUMMARY:
The purpose of this study is to compare two licensed influenza vaccines (Fluzone and Fluarix) in terms of the immune response elicited and the safety/ any symptoms that may occur for up to six months after vaccination.

DETAILED DESCRIPTION:
* Experimental design: multi-center, randomized (1:1), observer-blind, active-controlled study in 2 parallel groups with approximately:
* Study vaccine: full dose of Fluarix by IM administration.
* Control vaccine: full dose of Fluzone by IM administration.
* Two scheduled visits per subject at days 0 (visit 1) and 21(visit 2) with blood sample collected at each visit to evaluate the immune response. There will be a final contact with each subject 6 months after vaccination for safety follow up and study conclusion.
* Vaccination schedule: one IM injection at day 0.
* Type of study: Self contained.

ELIGIBILITY:
Inclusion Criteria:

* All adults 18 years and older.
* Subjects who the investigator believes can and will comply with the requirements of the protocol (e.g., return for follow-up visit and completion of the diary cards) should be enrolled in the study.
* Written informed consent obtained from the subject.
* If the subject is female, she must be of non-childbearing potential, i.e. either surgically sterilized or one year post-menopausal; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions .

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* History of hypersensitivity to a previous dose of influenza vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s) including egg, chicken protein, gelatine, formaldehyde, gentamicin sulphate, thimerosal or sodium deoxycholate.
* Acute disease at the time of enrollment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e. Oral temperature <37.5°C (99.5°F) / Axillary temperature <37.5°C (99.5°F)).
* History of Guillain Barré syndrome within 6 weeks of prior receipt of inactivated influenza virus vaccine.
* Pregnancy and lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1847 (Actual)
Dates: Start 2005-10; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Immunological non-inferiority (GMT & seroconversion rates) of Fluarix vs Fluzone 21 days post-vaccination in adults (18 yrs)

SECONDARY OUTCOMES:
Non-inferiority of Fluarix vs Fluzone 21 days post-vacc in elderly (>65 yrs)
Immuno comparison of Fluarix vs Fluzone post-vacc in immunologically -competent, -compromised, overall, stratified by age
Safety comparison (sol local, general & unsol AEs, SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (15):
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Campbell JD, Chambers CV, Brady RC, Caldwell MC, Bennett NL, Fourneau MA, Jain VK, Innis BL. Immunologic non-inferiority of a newly licensed inactivated trivalent influenza vaccine versus an established vaccine: a randomized study in US adults. Hum Vaccin. 2011 Jan 1;7(1):81-8. doi: 10.4161/hv.7.1.13553. Epub 2011 Jan 1. PMID 21285532
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104437 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104437 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104437 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104437 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104437 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104437 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104437 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register